CLINICAL TRIAL: NCT06649890
Title: A Randomized Control Trial Evaluating the Efficacy of Xperience™ Surgical Irrigation Solution Versus Dilute Povidone-Iodine in Preventing Surgical Site Infections and Improving Postoperative Outcomes in Implant-Based Breast Reconstruction
Brief Title: A Novel Surgical Irrigation Solution in Post-Mastectomy Reconstruction: Evaluating Xperience™
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24-0853
Record Dates: First submitted 2024-05-14; First posted 2024-10-21 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-06

CONDITIONS: Surgical Site Infection; Surgical Complication; Implant Infection; Implant Complication
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Xperience™ Advanced Surgical Irrigation (Experimental)
  Interventions: Device: Xperience™ Advanced Surgical Irrigation
- Dilute Povidone-Iodine (Active Comparator)
  Interventions: Device: Dilute Povidone-Iodine

INTERVENTIONS:
Device: Xperience™ Advanced Surgical Irrigation — Xperience™ solution will be applied twice during reconstruction procedures: first after achieving hemostasis and second just before implant introduction. The solution will be warmed to body temperature before use. Both tissue expanders/implants and mastectomy pockets will be soaked with Xperience™, using sterile syringes. A 1-minute dwell time with a total volume of 500 mL per mastectomy pocket will be employed, twice. Additionally, 500 mL of Xperience™ will be applied to implants before insertion, with a 5-minute dwell time. Excess solution will be suctioned throughout, and no rinsing will occur post-irrigation. Surgical site closure will follow standard procedures.
  Arms: Xperience™ Advanced Surgical Irrigation
Device: Dilute Povidone-Iodine — 5% dilute povidone-iodine solution will be prepared by mixing povidone-iodine solution and normal saline at the appropriate ratio. Both tissue expanders/implants and mastectomy pockets will be soaked with dilute povidone-iodine, using sterile syringes. A 1-minute dwell time with a total volume of 500 mL per mastectomy pocket will be employed, twice. Additionally, 500 mL of dilute povidone-iodine will be applied to implants before insertion, with a 5-minute dwell time. Excess solution will be suctioned throughout. Surgeon discretion will determine rinsing after irrigation. Surgical site closure will follow standard procedures.
  Other Names: Dilute Betadine
  Arms: Dilute Povidone-Iodine

SUMMARY:
Goal of the Clinical Trial:

The purpose of this clinical trial is to learn whether Xperience™ surgical irrigation solution is more effective than a standard dilute povidone-iodine solution in reducing surgical site infections (SSIs) following implant-based breast reconstruction in female patients, aged 18 and older. It will also assess the safety and overall surgical outcomes when using Xperience™ compared to povidone-iodine.

Main Questions the Study Aims to Answer:

* Does the use of Xperience™ decrease the incidence of surgical site infections compared to povidone-iodine?
* What are the differences in the rates of premature implant removal due to infection between patients treated with Xperience™ and those treated with povidone-iodine?
* Are there fewer post-surgical complications with Xperience™ compared to povidone-iodine?

Study Design:

Participants in this study will be randomly assigned to receive either Xperience™ or a dilute povidone-iodine solution during their bilateral implant-based breast reconstruction. Only the research team will know which irrgiation is given- the participant will not know.

Participant Will:

* Undergo the surgical procedure using one of the two irrigation solutions.
* Receive regular post-operative check-ups to monitor for signs of infection and other complications.
* Have data collected on any post-surgical complications, the necessity for early implant removal, and overall surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* Willing to comply with all study-related procedures
* Available for the duration of the study
* Participants undergoing double mastectomy surgery followed by one of the following: (1) Immediate reconstruction with tissue expander placement, (2) Delayed reconstruction with tissue expander or implant placement, (3) Immediate reconstruction with implant placement, (4) Second-stage reconstruction with tissue expander to implant exchange

Exclusion Criteria:

* Participants unable to participate in follow-up visits
* Participants undergoing unilateral mastectomy
* Tissue expanders placed by a surgeon outside of the UNC Chapel Hill Hospital System
* Undergoing autologous reconstruction
* Participant is unable to provide signed and dated informed consent
* Unwilling or unable to comply with all study-related procedures.
* Known history of sensitivity or allergic reaction to any of the components of the Xperience™ irrigation solution or dilute povidone-iodine irrigation
* Participant with any conditions that would be a contraindication to receiving surgery such as contraindications to general anesthesia
* Pregnant, planning to become pregnant or breast feeding participants
* Individuals providing informed consent with any mental impairment or condition that would make them unable to properly consent without use of legally authorized representative (LAR) or additional participant protections.
* Incarcerated participants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Surgical Site Infections | Within 90 days of implant/tissue expander placement, with the day of placement Day 0.
  Number of patients diagnosed with surgical site infections as per the diagnostic criteria outlined by the Centers for Disease Control National Healthcare Safety Network's 2024 Breast Surgery (BRST) Surgical Site Infection Criteria.

SECONDARY OUTCOMES:
Rate of Implant Explantation | Within 90 days of implant/tissue expander placement, with the day of placement Day 0.
  Number of patients who required non-elective implant explantation.
Rate of Non-Infectious Post-Surgical Complications | Within 90 days of implant/tissue expander placement, with the day of placement Day 0.
  Number of patients who experience the the following, but not limited to, post-surgical complications:
  * Delayed wound healing (superficial incisional dehiscence requiring serial dressing changes, office debridement and/or operative revision)
  * Hematoma
  * Seroma
  * Tissue expander leak/rupture
  * Tissue expander/Implant exposure/extrusion

CONTACTS AND LOCATIONS:
Overall Officials: Adeyemi Ogunleye, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No